CLINICAL TRIAL: NCT05494606
Title: Prospective Real World Study Of Upadacitinib in Ulcerative Colitis (PROFUNDUS)
Brief Title: An Observational Study to Assess Change in Disease Activity and Adverse Events of Upadacitinib in Adult Participants With Moderate to Severe Ulcerative Colitis (UC) in Real-World Practice
Acronym: PROFUNDUS
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-921
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Upadacitinib; PROFUNDUS; RINVOQ
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving upadacitinib: Participants receiving upadacitinib for moderate to severe Ulcerative colitis (UC) in real-world practice.

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic, inflammatory disease affecting the colon. Participants with UC have mucosal inflammation starting in the rectum that can extend continuously to proximal segments of the colon. This study will assess how safe and effective upadacitinib is in treating adult participants with moderate to severe ulcerative colitis (UC). Adverse events and change in disease activity will be assessed.

Upadacitinib is a drug approved for the treatment of Ulcerative colitis (UC). All study participants will receive upadacitinib as prescribed by their study doctor in accordance with approved local label. Approximately 1000 adult participants will be enrolled worldwide.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 3 years.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate to severe Ulcerative colitis (UC).
* Participants initiating upadacitinib at the clinician's discretion as part of their routine clinical care; the decision to administer upadacitinib must be made prior to and independent of recruitment into the study.
* Participants prescribed upadacitinib in accordance with the approved local label.
* Participants able to understand and communicate with the investigator and comply with the requirements of the study.
* Participants willing to continue with study documentation after cessation of upadacitinib.
* Participants willing and able to participate in the collection of patient-reported data via cloud based mobile application using the provided smart device (iPhone).

Exclusion Criteria:

* Participants with any contraindication to upadacitinib.
* Participants previously exposed to upadacitinib in a clinical trial.
* Participants currently participating in interventional research (not including noninterventional study, postmarketing observational study (PMOS), or registry participation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active Ulcerative colitis (UC)
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Median Time to Achieve the First Clinical Response (CR) per Partial Adapted Mayo Score | Up to approximately week 156
  The first clinical response (CR) per partial adapted mayo score is defined as a decrease from baseline in partial adapted mayo score ≥ 1 point and ≥ 30%, plus a decrease from baseline in the rectal bleeding score [RBS] ≥ 1 or absolute RBS ≤ 1. Median time to achieve the first CR per partial adapted mayo score will be reported
Percentage of Participants Achieving Clinical Response (CR) per Partial Adapted Mayo Score Among those who Achieved CR at Completion of Upadacitinib Induction (either at Week 8 or at Week 16) | Week 52
  Clinical response (CR) per partial adapted mayo score is defined as a decrease from baseline in partial adapted mayo score ≥ 1 point and ≥ 30%, plus a decrease from baseline in the rectal bleeding score [RBS] ≥ 1 or absolute RBS ≤ 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (153):
- Argentina (3):
  - Gedyt /ID# 249611, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires /ID# 249605, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 249612, Córdoba
- Australia (5):
  - Blacktown Hospital /ID# 248354, Blacktown, New South Wales
  - Nepean Hospital /ID# 248351, Kingswood, New South Wales
  - Coral Sea Clinical Research institute /ID# 248352, North Mackay, Queensland
  - Austin Health /ID# 249133, Heidelberg, Victoria
  - The Royal Melbourne Hospital /ID# 248353, Parkville, Victoria
- Canada (16):
  - University of Calgary /ID# 259183, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institution /ID# 251463, Edmonton, Alberta
  - Dr. J Siffledeen Profess Pract /ID# 256903, Edmonton, Alberta
  - Six08 Gastroenterology /ID# 259452, Lethbridge, Alberta
  - Dr. Sundeep Singh, Inc /ID# 251471, Kelowna, British Columbia
  - The Moncton Hospital /ID# 257337, Moncton, New Brunswick
  - Barrie GI Associates /ID# 264978, Barrie, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 256819, Hamilton, Ontario
  - London Health Sciences Center- University Hospital /ID# 258472, London, Ontario
  - West GTA Endoscopy /ID# 263221, Mississauga, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 256826, North Bay, Ontario
  - Toronto Immune and Digestive Health Institute Inc /ID# 256827, North York, Ontario
  - Toronto Digestive Disease Associates /ID# 258914, Vaughan, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 260528, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 258470, Montreal, Quebec
  - Diex Recherche Québec /ID# 262796, Québec, Quebec
- Czechia (5):
  - Iscare Klinické Centrum /ID# 259811, Prague, Praha 9
  - SurGal Clinic /ID# 259809, Brno, South Moravian
  - Nemocnice Ceske Budejovice a.s. /ID# 259810, České Budějovice
  - Fakultni nemocnice Kralovske Vinohrady /ID# 261535, Prague
  - Fakultni Thomayerova nemocnice /ID# 261626, Prague
- France (31):
  - Chu de Nice-Hopital L'Archet Ii /Id# 251938, Nice, Alpes-Maritimes
  - APHM - Hopital Nord /ID# 252049, Marseille, Bouches-du-Rhone
  - CHU de Besancon - Jean Minjoz /ID# 252966, Besançon, Doubs
  - CHU NIMES - Hopital Caremeau /ID# 254790, Nîmes, Gard
  - Hôpitaux Civils de Colmar - Hôpital Pasteur /ID# 252496, Colmar, Grand Est
  - CHU Toulouse - Hopital Rangueil /ID# 251879, Toulouse, Haute-Garonne
  - CHU Montpellier - Hopital Saint Eloi /ID# 252041, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 251937, La Tronche, Isere
  - Clinique Santé Atlantique /ID# 252581, Saint-Herblain, Loire-Atlantique
  - CHU Reims - Hôpital Robert Debre /ID# 252017, Reims, Marne
  - CHRU Lille - Hopital Claude Huriez /ID# 251971, Lille, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 251972, Créteil, Paris
  - AP-HP - Hopital Bicetre /ID# 252329, Le Kremlin-Bicêtre, Paris
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord /ID# 252265, St-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier D'Avignon /ID# 252657, Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Cote Basque /ID# 252358, Bayonne, Pyrenees-Atlantiques
  - HCL - Hopital Lyon Sud /ID# 252093, Pierre-Bénite, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 252103, Amiens, Somme
  - Clinique de l'Europe /ID# 251851, Amiens, Somme
  - Ch Bethune - Beuvry /Id# 252233, Béthune
  - Pole Sante Saint-Jean /ID# 252235, Cagnes-sur-Mer
  - CH Annecy Genevois - Site Annecy /ID# 253010, Epagny Metz Tessy
  - GHI Le Raincy - Montfermeil /ID# 252733, Montfermeil
  - Clinique Jules Verne /ID# 251969, Nantes
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 252125, Orléans
  - Institut Mutualiste Montsouris /ID# 251849, Paris
  - CHRU Pontchaillou /ID# 252015, Rennes
  - Centres des maladies de l'appareil digestif /ID# 252283, Strasbourg
  - Clinique Pasteur /ID# 251893, Toulouse
  - Hôpital Schuman /ID# 252995, Vantoux
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 252565, Neuilly-sur-Seine, Île-de-France Region
- Germany (32):
  - Medizinisches Versorgunszentrum Dachau /ID# 257231, Dachau, Bavaria
  - Praxis Dres. Hurst/Simonis /ID# 255159, Darmstadt, Hesse
  - Interdisziplinaeres Crohn Colitis Zentrum /ID# 252224, Frankfurt am Main, Hesse
  - Markus Krankenhaus /ID# 260648, Frankfurt am Main, Hesse
  - Gastroenterologie Opernstrasse Private Practice - Dr. Falk & Krause & Kuhn /ID# 252076, Kassel, Hesse
  - Magen-Darm-Zentrum-Remscheid /ID# 250339, Remscheid, North Rhine-Westphalia
  - Duplicate_St. Marien- und Annastiftskrankenhaus /ID# 255158, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 251824, Saarbrücken, Saarland
  - Internistische Gemienschaftspraxis fuer Verdauungs- und Stoffwechselerkrankungen /ID# 250873, Leipzig, Saxony
  - Private Practice - Dr. Thomas Zeisler /ID# 250126, Halle, Saxony-Anhalt
  - Praxis S. Tetzlaff /ID# 248263, Buedelsdorf, Schleswig-Holstein
  - Thurman/Bethge /ID# 248305, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 251273, Lübeck, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 250749, Lübeck, Schleswig-Holstein
  - Dr. Bernd Adami /ID# 248123, Alzey
  - Dr. Heil /ID# 248273, Andernach
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 248979, Berlin
  - Praxis Dr. Michael Mross /ID# 248272, Berlin
  - Krankenhaus Waldfriede /ID# 248307, Berlin-Zehlendorf
  - Praxis Dr. Lukas Buendgens & Dr. Burkhard Buendgens /ID# 254873, Eschweiler
  - Dres. Bauer/Doerflinger /ID# 252107, Freiburg im Breisgau
  - Dres. Behrens/Fechner/Streudel /ID# 250872, Halle
  - Miamedes Hausarztpraxis Altona /ID# 260064, Hamburg
  - Medizinische Hochschule Hannover /ID# 257454, Hanover
  - GSGH Gastroenterologische Studiengesellschaft Herne GbR /ID# 250262, Herne
  - Dres. Breitschwerdt/Glas/Gurtler /ID# 251192, Leipzig
  - Bettenworth & Partner /ID# 248977, Münster
  - Gastro Campus Research GbR /ID# 249867, Münster
  - Gastro.Praxis am Meerbachbogen /ID# 251856, Nienburg
  - Praxis Dres Brendel /ID# 250559, Nuremberg
  - Schwerpunktpraxis Gastroenterologie Dr. Ingomar Scheller /ID# 250581, Remscheid
  - Praxis Dr. Kempelmann /ID# 257748, Tostedt
- Greece (7):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 260787, Athens, Attica
  - Alexandra General Hospital /ID# 260786, Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" /ID# 250794, Nikaia, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 259869, Heraklion, Crete
  - University General Hospital of Alexandroupoli /ID# 270159, Alexandroupoli, Evros
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 259870, Athens
  - General Hospital of Thessaloniki Hippokrateio /ID# 260785, Thessaloniki
- Ireland (3):
  - Connolly Hospital Blanchardstown /ID# 252190, Abbotstown, Dublin
  - St Vincent's University Hospital /ID# 251855, Elm Park, Dublin
  - University Hospital Galway /ID# 253427, Galway
- Israel (5):
  - Shamir Medical Center /ID# 256885, Beer Ya'akov, Central District
  - Rambam Health Care Campus /ID# 249884, Haifa, H_efa
  - Soroka University Medical Center /ID# 249885, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 250562, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 249474, Petah Tikva
- Italy (10):
  - Ente Ospedaliero Specializzato in Gastroenterologia Saverio de Bellis - IRCCS /ID# 261600, Castellana Grotte, Bari
  - IRCCS Istituto Clinico Humanitas /ID# 260801, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 261058, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 260802, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 260811, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 260946, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 261116, Negrar, Verona
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 260812, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 261052, Palermo
  - Azienda Ospedaliero Universitaria Pisana /ID# 261126, Pisa
- Mubarak Hospital /ID# 252026, Hawalli, Kuwait
- Portugal (8):
  - Hospital Central da Madeira, Hospital Dr. Nélio Mendonça /ID# 271710, Funchal, Madeira
  - Hospital Garcia de Orta /ID# 264420, Almada, Setúbal District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital Faro /ID# 260517, Faro
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz /ID# 260524, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 258759, Lisbon
  - Unidade Local de Saude de Loures-Odivelas, EPE /ID# 272785, Loures
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 260038, Porto
  - Centro Hosp de Tondela-Viseu /ID# 258760, Viseu
- Hamad Medical Corporation /ID# 253823, Zone 51, Baladīyat ar Rayyān, Qatar
- Voronezh Regional Clinical Hospital #1 /ID# 249932, Voronezh, Russia
- Spain (11):
  - Hospital Universitari de Bellvitge /ID# 263932, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Parc Tauli /ID# 263931, Sabadell, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín /ID# 263929, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de Cabueñes /ID# 263930, Gijón, Principality of Asturias
  - Hospital Universitario de Canarias /ID# 264214, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Virgen Macarena /ID# 263924, Seville, Sevilla
  - Hospital Universitario Virgen del Rocio /ID# 263926, Seville, Sevilla
  - Hospital Galdakao-Usansolo /ID# 263925, Galdakao, Vizcaya
  - Hospital Universitario Torrecárdenas /ID# 264202, Almería
  - Hospital Juan Ramón Jiménez /ID# 267702, Huelva
  - Hospital Universitario de Salamanca /ID# 264207, Salamanca
- United Arab Emirates (2):
  - Burjeel Day Surgery Center /ID# 252030, Abu Dhabi
  - Cleveland Clinic Abu Dhabi /ID# 252038, Abu Dhabi
- United Kingdom (12):
  - Royal Devon & Exeter Hospital /ID# 252734, Exeter, Devon
  - Hull University Teaching Hospitals NHS Trust /ID# 253988, Hull, East Riding Of Yorkshire
  - Hampshire Hospitals NHS Foundation Trust /ID# 261416, Basingstoke, Essex
  - Northern Care Alliance NHS Foundation Trust /ID# 253993, Bury, Lancashire
  - Kettering General Hospital NHS Foundation Trust /ID# 255263, Kettering, Northamptonshire
  - Nottingham City Hospital /ID# 255270, Nottingham, Nottinghamshire
  - Oxford University Hospitals - John Radcliffe Hospital /ID# 265343, Oxford, Oxfordshire
  - Ulster Hospital - South Eastern Health & Social Care Trust /ID# 255265, Belfast
  - Liverpool University Hospitals NHS Foundation Trust /ID# 253989, Liverpool
  - Barts Health NHS Trust /ID# 252735, London
  - St George's University Hospitals NHS Foundation Trust /ID# 255271, Tooting
  - New Cross Hospital /ID# 266364, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=P22-921